CLINICAL TRIAL: NCT03557242
Title: Strategies to Prevent Transcatheter Heart Valve Dysfunction in Low Risk Transcatheter Aortic Valve Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LRT 2.0
Record Dates: First submitted 2018-05-29; First posted 2018-06-14 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Warfarin; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Warfarin plus Aspirin (Other): 100 subjects will be randomized electronically through the Electronic Data Capture System in a 1:1 fashion to warfarin plus low dose aspirin for 30-45 days
  Interventions: Device: TAVR; Other: Warfarin plus Aspirin
- Aspirin Monotherapy (Other): 100 subjects will be randomized electronically through the Electronic Data Capture System in a 1:1 fashion to low dose aspirin monotherapy for 30-45 days
  Interventions: Device: TAVR; Other: Aspirin Only
- Registry Arm (Other): Upto an additional 100 subjects with preexisting indication for anti coagulation (e.g. atrial fibrillation, deep venous thrombosis, pulmonary embolism) or who are not eligible for randomization after TAVR due to development of a new indication for anti coagulation will be enrolled in the registry arm of the study.
  Interventions: Device: TAVR

INTERVENTIONS:
Device: TAVR — Transcatheter Aortic Valve Replacement
Other: Warfarin plus Aspirin — Subjects randomized to this arm will receive Warfarin plus aspirin for 30- 45 days post TAVR
  Arms: Warfarin plus Aspirin
Other: Aspirin Only — Subjects randomized to this arm will receive aspirin only post TAVR
  Arms: Aspirin Monotherapy

SUMMARY:
100 subjects in the each of the treatment arms of the study (total 200 treatment arm subjects) and up to 100 subjects in the registry arm of the study.

DETAILED DESCRIPTION:
This study aims to examine the optimal anticoagulation/antiplatelet regimen in low risk patients undergoing TAVR. The prospective randomized controlled arm of this study will assess the utility of short-term oral anticoagulation with warfarin compared to antiplatelet therapy alone after TAVR in low risk patients to reduce the incidence of structural valve deterioration manifest as clinical events, increased aortic valve gradients or transvalvular regurgitation, or subclinical leaflet thrombosis. Low risk subjects with symptomatic severe aortic stenosis will be enrolled to undergo TAVR. Following TAVR, subjects will be randomized to receive warfarin plus low dose Aspirin or low dose Aspirin monotherapy for 30-45 days. Subjects with other indications for anticoagulation (e.g. AF, DVT or PE) will not be randomized and instead will be followed in a separate registry arm. Baseline demographic, clinical, non-invasive imaging (echocardiography and CT), TAVR procedural details, clinical follow up data will be prospectively collected for all subjects. Echocardiography and contrast-enhanced 4D cardiac CT will be performed in all subjects between 30-45 days after TAVR to evaluate for evidence of structural valve deterioration.

This multicenter prospective randomized study will enroll 200 consecutive low risk subjects with symptomatic severe aortic stenosis into the treatment arms of the study. Up to 100 additional subjects with a pre-existing indication for anticoagulation (e.g. atrial fibrillation, deep venous thrombosis or pulmonary embolism) or who are not eligible for randomization after TAVR due to development of a new indication for anticoagulation will be enrolled into the registry arm of the study.

Inclusion of this registry arm will ensure that the secondary objective pooled analysis of patient level data from this study and the Low Risk TAVR (LRT) study, truly represents an all-comers cohort of low risk patients undergoing TAVR, and does not exclude a significant subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Severe, degenerative AS, defined as:
* Mean aortic valve gradient ≥40 mm Hg OR Vmax ≥4 m/sec AND
* Calculated aortic valve area ≤1.0 cm2 OR aortic valve area index ≤0.6 cm2/m2
* Symptomatic AS, defined as a history of at least one of the following:
* Dyspnea that qualifies at New York Heart Association (NYHA) class II or greater
* Angina pectoris
* Cardiac syncope
* The Heart Team agrees that the patient is low-risk, quantified by an estimated risk of death ≤3% by the calculated STS score for operative mortality at 30 days; AND agrees that SAVR would be an appropriate therapy if offered
* A surgeon who is experienced in Surgical Aortic Valve Replacement (SAVR) has spoken with the patient in person and stipulates that the patient understands his/her alternatives for FDA approved therapy, including open heart surgery to replace their aortic valve
* The institutional Heart Team determines that transfemoral TAVR is appropriate
* Aortic valve anatomy and dimensions suitable for TAVR using a commercially available valve
* Iliofemoral artery anatomy and dimensions suitable for transfemoral TAVR using a commercially available valve and delivery system
* Procedure status is elective
* Expected survival is at least 24 months

Exclusion Criteria:

* Subject unable or unwilling to give informed consent
* Concomitant disease of another heart valve or the aorta that requires either transcatheter or surgical intervention
* Any condition that is considered a contraindication for placement of a bioprosthetic aortic valve (e.g. patient requires a mechanical aortic valve)
* Aortic stenosis secondary to a bicuspid aortic valve
* Prior bioprosthetic surgical aortic valve replacement
* Mechanical heart valve in another position
* End-stage renal disease requiring hemodialysis or peritoneal dialysis, or a creatinine clearance <20 cc/min
* Left ventricular ejection fraction <20%
* Recent (<6 months) history of stroke
* Symptomatic carotid or vertebral artery disease, or recent (<6 weeks) surgical or endovascular treatment of carotid stenosis
* Any contraindication to oral antiplatelet or anticoagulation therapy following the procedure, including recent or ongoing bleeding, or HASBLED score >3 (Table 2 - HASBLED scoring system)
* Severe coronary artery disease that is unrevascularized
* Recent (<30 days) acute myocardial infarction
* Patient cannot undergo transfemoral TAVR for anatomic reasons (as determined by supplemental imaging studies); this would include inadequate size of iliofemoral access vessels or an aortic annulus size that is not accommodated by the commercially available valves
* Any comorbidity not captured by the STS score that would make SAVR high risk, as determined by a cardiothoracic surgeon who is a member of the heart team; this includes:
* Porcelain or severely atherosclerotic aorta
* Frailty
* Hostile chest
* Internal mammary artery or other conduit either crosses midline of sternum or is adherent to sternum
* Severe pulmonary hypertension (PA systolic pressure > 2/3 of systemic pressure)
* Severe right ventricular dysfunction
* Ongoing sepsis or infective endocarditis
* Severe chronic obstructive pulmonary disease, as demonstrated by forced expiratory volume (FEV1) <750 cc
* Liver failure with Childs class C or D
* Pre-procedure shock, inotropes, mechanical assist device, or cardiac arrest
* Pregnancy or intent to become pregnant prior to completion of all protocol follow-up procedures
* Known allergy to warfarin or aspirin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
All Cause Mortality | 30 days
All Stroke | 30 days
  disabling and non-disabling, ischemic, hemorrhagic
Life-threatening and Major Bleeding | 30 days
Major Vascular Complications | 30 Days
Hospitalizations for valve-related symptoms or worsening congestive heart failure | 30 days
Hypoattenuated leaflet thickening (HALT) | 30 days
At least moderately restricted leaflet motion (RELM) | 30 days
Hemodynamic dysfunction | 30 Days
  (mean aortic valve gradient ≥20 mm Hg, AND/OR EOA ≤1.0 cm2 AND/OR DVI<0. 35, AND/OR moderate or severe prosthetic valve regurgitation)

SECONDARY OUTCOMES:
VARC-2 device success: | 1 year
  * Absence of procedural mortality AND
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location AND
  * Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient<20 mm Hg or peak velocity<3 m/s, AND no moderate or severe prosthetic valve regurgitation)
All-cause mortality | 1 year
All stroke | 1 year
  (disabling and non-disabling, ischemic and hemorrhagic)
Life-threatening and major bleeding | 1 year
Major vascular complications | 1 year
Hospitalizations for valve-related symptoms or worsening congestive heart failure | 1 year
Acute kidney injury | 1 year
Pacemaker implantation | 1 year
Endocarditis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ron S Waksman, MD, Principal Investigator — MedStar Cardiovascular Research Network
Locations (7):
- United States (7):
  - Foundation for Cardiovascular Medicine, San Diego, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - The Valley Hospital, Ridgewood, New Jersey
  - Stony Brook Hospital, Stony Brook, New York
  - St. John Health System, Tulsa, Oklahoma
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Henrico Doctors' Hospital, Richmond, Virginia

REFERENCES:
- [Derived] Bhogal S, Waksman R, Shea C, Zhang C, Gordon P, Ehsan A, Wilson SR, Levitt R, Parikh P, Bilfinger T, Hanna N, Buchbinder M, Asch FM, Weissman G, Ben-Dor I, Shults CC, Ali S, Garcia-Garcia HM, Satler LF, Rogers T. Self-expanding and balloon-expandable valves in low risk TAVR patients. Int J Cardiol. 2024 Jan 15;395:131431. doi: 10.1016/j.ijcard.2023.131431. Epub 2023 Oct 12. PMID 37832606
- [Derived] Medranda GA, Soria Jimenez CE, Torguson R, Case BC, Forrestal BJ, Ali SW, Shea C, Zhang C, Wang JC, Gordon P, Ehsan A, Wilson SR, Levitt R, Parikh P, Bilfinger T, Hanna N, Buchbinder M, Asch FM, Weissman G, Shults CC, Garcia-Garcia HM, Ben-Dor I, Satler LF, Waksman R, Rogers T. Lifetime management of patients with symptomatic severe aortic stenosis: a computed tomography simulation study. EuroIntervention. 2022 Aug 5;18(5):e407-e416. doi: 10.4244/EIJ-D-21-01091. PMID 35321859
- [Derived] Rogers T, Shults C, Torguson R, Shea C, Parikh P, Bilfinger T, Cocke T, Brizzio ME, Levitt R, Hahn C, Hanna N, Comas G, Mahoney P, Newton J, Buchbinder M, Moreno R, Zhang C, Craig P, Asch FM, Weissman G, Garcia-Garcia HM, Ben-Dor I, Satler LF, Waksman R. Randomized Trial of Aspirin Versus Warfarin After Transcatheter Aortic Valve Replacement in Low-Risk Patients. Circ Cardiovasc Interv. 2021 Jan;14(1):e009983. doi: 10.1161/CIRCINTERVENTIONS.120.009983. Epub 2021 Jan 11. PMID 33423540